CLINICAL TRIAL: NCT06886451
Title: Prevention of Vomiting in Pediatric Oncology Inpatients Using Machine Learning
Brief Title: Vomiting Prevention in Children With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lillian Sung, Chief Clinical Data Scientist, Paediatric Oncologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3373
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Chemotherapy Induced Nausea and Vomiting; Quality of Life (QOL); Pediatric Cancer
Keywords: Vomiting; Machine learning; Quality of life; Pediatric oncology
MeSH Terms: conditions — Vomiting; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ML model (Experimental): ML model to predict the risk of vomiting within the next 96 hours.
  Interventions: Other: ML-based intervention

INTERVENTIONS:
Other: ML-based intervention — For each patient, a ML model will predict the risk of vomiting within the next 96 hours. Patients will then receive care pathway-consistent interventions based on the ML model predictions.
  Other Names: Machine learning model

SUMMARY:
The goal of this single arm trial is to learn if a machine learning (ML) model predicting the risk of vomiting within the next 96 hours will impact vomiting outcomes in inpatient cancer pediatric patients.

The main questions it aims to answer are whether an ML model predicting the risk of vomiting within the next 96 hours will:

Primary

1. Reduce the proportion with any vomiting within the 96-hour window

Secondary

1. Reduce the number of vomiting episodes
2. Increase the proportion receiving care pathway-consistent care
3. Impact on number of administrations and costs of antiemetic medications

Newly admitted participants will have a ML model predict the risk of vomiting within the next 96 hours according to their medical admission information. The prediction will be made at 8:30 AM following admission. Pharmacists will be charged with bringing information about patients' vomiting risk to the attention of the medical team and implementing interventions.

DETAILED DESCRIPTION:
Vomiting is one of the most common complications of cancer therapies in pediatric patients, with substantial negative impacts on quality of life. Vomiting can also reduce oral intake, worsen nutritional status and lead to hospitalization. Thus, efforts to control vomiting are crucial. The ability to predict which patients are most likely to vomit is limited; machine learning (ML) is a promising approach. Preliminary work completed for this study includes development of an enterprise data warehouse sourced from Epic suitable for ML named SickKids Enterprise-wide Data in Azure Repository (SEDAR) and validation of vomiting outcomes in SEDAR. Next, a standardized process for model training, evaluation and deployment was conducted by the study team. This was implemented to train a retrospective model to predict vomiting (0-96 hours post prediction time), which demonstrated satisfactory performance during a prospective silent trial. The care pathway and patient-specific report to facilitate clinical care based on a positive prediction has also been created by the study team, expending on a previously developed antiemetic care pathway based on clinical practice guidelines. The patient-specific report lists each patient's risk of vomiting (0-96 hours post prediction time), vomiting prior to prediction time, planned chemotherapy or procedures, current antiemetic orders and history of vomiting with the most recent admission.

For model deployment, pharmacists will be charged with bringing information about patients' vomiting risk to the attention of the medical team and implementing care pathway-consistent interventions. Pharmacists will receive a list of high-risk patients and the developed tools (care pathway and patient-specific report) each morning. Outcomes will be evaluated for a one-year period pre- and post-deployment. Primary outcome will be any vomiting within the 96-hour period post prediction time. Secondary outcomes will be the number of vomiting episodes within the 96-hour period, care pathway-consistent care, antiemetic administrations and antiemetic costs.

The study team includes pediatric pharmacists, pediatric oncologists and experts in machine learning, clinical epidemiology, implementation sciences, care pathway development and biostatistics.

Vomiting is one of the most distressing aspects of cancer therapy and, with current approaches, medical management is failing a substantial number of patients. This work will contribute to precision medicine by identifying patients with the highest need for individualized review and therapy optimization. This effort is anticipated to improve the quality of care and quality of life for pediatric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients admitted to the oncology service at SickKids

Exclusion Criteria:

* Pediatric patients admitted to the oncology service at SickKids that are discharged prior to prediction time

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1332 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-03-18 (Estimated); Study Completion 2027-03-18 (Estimated)

PRIMARY OUTCOMES:
Vomiting post prediction time | 0-96 hours post prediction time
  The primary outcome will be any vomiting (a binary variable) 0-96 hours post prediction time. In the SickKids EHR, vomiting is described in the flowsheets by emesis volume, emesis count, emesis amount description, emesis color/appearance, and any vomiting/retching/gagging. Multiple descriptors can be used at a specific time stamp but no one descriptor is used consistently. Thus, the best measure of vomiting is a binary variable (yes/no) where yes represents any vomiting entry within the 96-hour window. Vomiting determination using this approach was validated. In a retrospective assessment, patients who received etoposide, ifosfamide or treosulfan were identified and 60 patients were randomly selected with stratification by age and HCT status. (Patel P et al, 2023)

SECONDARY OUTCOMES:
Number of episodes of vomiting | 0-96 hours post prediction time
  The number of episodes of vomiting will be determined by counting the number of distinct time stamps with any vomiting description.
Care pathway-consistent care | 0-96 hours post prediction time
  Care pathway-consistent care will be measured as a binary outcome (yes/no).
Number of antiemetic administrations | 0-96 hours post prediction time
  All antiemetic administrations within the 96-hour window will be counted. The total number of administrations overall and by specific antiemetic agent will be tabulated.
Antiemetic costs | 0-96 hours post prediction time
  Medication costs are available in SEDAR. The total costs of antiemetics per kg overall and by specific antiemetic agent will be tabulated.

OTHER OUTCOMES:
Number of SEDAR Predictions and Interventions | 0-96 hours post prediction time
  The number of times notes in SEDAR refer to the predictions and interventions to address them including antiemetic modifications during the prediction window will be descriptively reported. The role of the note writer will be documented (such as pharmacist or fellow).

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, PhD, Principal Investigator — The Hospital for Sick Children; Lee Dupuis, RPh, PhD, Principal Investigator — The Hospital for Sick Children; Priya Patel, PharmD, Principal Investigator — The Hospital for Sick Children; Adam Yan, MD, MBI, Principal Investigator — The Hospital for Sick Children; Lawrence Guo, PhD, Principal Investigator — The Hospital for Sick Children; Santiago Arciniegas, MSc, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel P, Robinson PD, Phillips R, Baggott C, Devine K, Gibson P, Guilcher GMT, Holdsworth MT, Neumann E, Orsey AD, Spinelli D, Thackray J, van de Wetering M, Cabral S, Sung L, Dupuis LL. Treatment of breakthrough and prevention of refractory chemotherapy-induced nausea and vomiting in pediatric cancer patients: Clinical practice guideline update. Pediatr Blood Cancer. 2023 Aug;70(8):e30395. doi: 10.1002/pbc.30395. Epub 2023 May 13. PMID 37178438